CLINICAL TRIAL: NCT03297775
Title: Rheumatoid Arthritis Patients at Risk for Interstitial Lung Disease
Acronym: RAPID
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1097
Record Dates: First submitted 2017-09-19; First posted 2017-09-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: Rheumatoid Arthritis; RA; Interstitial Lung Disease; ILD; lung disease; connective tissue disease; CTD; idiopathic pulmonary fibrosis; IPF; airways disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial; Lung Diseases; Connective Tissue Diseases; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — The following bio-specimens will be collected at baseline and at 3-5 years follow-up:
  * DNA (baseline only)
  * RNA
  * PBMC, Serum, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA with Sub-clinical ILD: Subjects will be followed annually until study closure.
  Assessments are as follows:
  1. Clinical (Annual): Demographics, health-related behaviors, co-morbidities, medications, respiratory symptoms, rheumatologic assessment, quality of life
  2. Physiologic (3-5 yrs FU): Lung function on Pulmonary Function Test (PFT)
  3. Radiologic (3-5 yrs FU): HRCT scan of chest
  4. Genetic (3-5 yrs FU): Blood sample collection for RNA
  5. Biologic (3-5 yrs FU): Blood sample collection for other blood markers
- RA with No-ILD: Subjects will be followed annually until study closure.
  Assessments are as follows:
  1. Clinical (Annual): Demographics, health-related behaviors, co-morbidities, medications, respiratory symptoms, rheumatologic assessment, quality of life
  2. Physiologic (3-5 yrs FU): Lung function on Pulmonary Function Test (PFT)
  3. Radiologic (3-5 yrs FU): HRCT scan of chest
  4. Genetic (3-5 yrs FU): Blood sample collection for RNA
  5. Biologic (3-5 yrs FU): Blood sample collection for other blood markers
  Note: Certain follow-up procedures may not occur for every subject and will be determined by the research team.

SUMMARY:
The overall goal of this study is to define the phenotype of Interstitial Lung Disease (ILD), and identify factors that predict radiologic progression in those with subclinical RA-ILD, in patients with rheumatoid arthritis (RA). The investigators hypothesize that there are common core elements (e.g. clinical features, genetic variants, and/or biologic markers) between other forms of ILD (e.g. idiopathic pulmonary fibrosis, IPF) and subclinical RA-ILD that places individuals at risk for the development of lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 45years old
2. Diagnosis of RA using the 2010 American College of Rheumatology (ACR) criteria

Exclusion Criteria:

1. Inability to give informed consent
2. Pregnant women
3. History of interstitial lung disease
4. Evidence of other causes of diffuse parenchymal lung disease such as infection, drug toxicity, other autoimmune processes, etc.
5. Subjects over the age of 90 years old or less than 45 years old

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are selected for participation in the study because they have an active diagnosis of rheumatoid arthritis and are at risk for the development of lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Presence of interstitial lung disease on high resolution CT (HRCT) chest imaging | 3-5 years
  HRCT scans of the chest will be interpreted by two radiologists and the presence or absence of interstitial lung abnormality will be recorded. When present, abnormalities will be categorized as absent, equivocal, non-fibrotic, or fibrotic, and the extent of any reticular abnormalities will be graded on an 11-point scale (0, 1-10%, 11-20%, etc.). Additionally, the presence or absence of airway disease, centrilobular thickening, mosaic attenuation, and air trapping will be recorded.

SECONDARY OUTCOMES:
Progression of lung disease over time | 3-5 Years
  Radiologic progression of lung disease will be determined through a comparison of baseline HRCT chest findings to follow-up HRCT chest findings at the 3-5 year follow-up benchmark. Similar to baseline, follow-up HRCT scans of the chest will be interpreted by 2 different radiologists. Quantitative radiologic progression will be defined as ≥ 10% increase in fibrotic changes from baseline to follow-up - additionally, the percent reticular change, percent honeycomb change, and percent traction bronchiectasis on the follow-up scan will be quantified and recorded.
  Radiologic findings of progression will be used in correlation with other clinical features to determine the clinical relevance of the change. The clinical features include - change in cough, change in dyspnea (as measured by UCSD shortness of breath questionnaire), change in FVC percent predicted value, the development of established RA-ILD, or respiratory-related death, over the same time period.
Impact of subclinical RA-ILD on health-related quality of life in RA | 3-5 Years
  The impact of subclinical RA-ILD on health-related quality of life will be measured using subjective patient questionnaires that will be completed at both baseline and follow-up. These questionnaires include - SF-36, St. George Respiratory Questionnaire, and Multi-Dimensional Health Assessment Questionnaire.
Outcome of airways disease | 3-5 Years
  Clinical outcomes will be measured through respiratory assessment (physical exam), changes is dyspnea (based on the University of California San Diego shortness of breath questionnaire), changes in FVC percent predicted values (based on pulmonary function testing), increase in cough (determined using a visual analog scale, where 10 is the worst cough and 0 is no cough), and development of RA-ILD requiring treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce S Lee, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No